CLINICAL TRIAL: NCT06744816
Title: Exploring the Benefit of Topical Capsaicin in Treating Pain From Chemo-induced Peripheral Neuropathy: a Longitudinal Single Center Pilot Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Averitas Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1601; NCI-2024-10413 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Qutenza Patch (Topical Capsaicin) (Experimental): Up to 4 topical capsaicin patches will be applied on your feet for 30 minutes.
  Interventions: Drug: Qutenza Patch

INTERVENTIONS:
Drug: Qutenza Patch — Given topical

SUMMARY:
To learn if topical capsaicin can help relieve pain from CIPN and improve gait (the pattern of walking) in patients.

DETAILED DESCRIPTION:
Primary Objectives

• To assess changes in Gait (specifically looking at velocity) before and after use of topical capsaicin.

Secondary Objectives

* To assess Pain intensity numerical rating scale (NRS) scores in chemotherapy induced peripheral neuropathy (CIPN) participants before and after use of capsaicin 8% topical patch.
* To assess changes in quantitative sensory testing (QST) before and after use of topical capsaicin.
* To assess skin punch biopsy to compare the integrity of epidermal nerve fibers and Meissner's corpuscles (MC) in CIPN patients before and after use of topical capsaicin (optional).
* To assess pain tumor related neuropathy assessment scale (TNAS) before and after topical capsaicin
* To assess pain interference using the Brief Pain Inventory (BPI), before and after topical capsaicin
* To assess Patient Global Impression of Change (PGIC)
* To assess the rate of adverse events and tolerability of topical capsaicin as reported by participants

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with pain of the lower extremity from chronic (>90 days duration) CIPN (due to either vinca alkaloids, taxanes, bortezomib, thalidomide, platinum-based compounds), seen at MD Anderson Cancer Center
* Participants reporting baseline pain ≥ 4 (0-10 scale, NRS)
* Participants age 18+
* Participants who have completed chemotherapy within the last year at the time of enrollment.

Exclusion Criteria:

* Participants with cognitive dysfunction
* Participants with recent history (<6 months) of drug or alcohol abuse
* Participants with open skin lesion or undergoing antibiotic therapy for local for systemic infection
* Participants with allergies to capsaicin or adhesives
* Pregnant participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AE)s | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Saba Javed, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org